CLINICAL TRIAL: NCT03561714
Title: Cardiometabolic Care-team Integration in Primary Care Improves Outcomes in Diabetes: a Pragmatic, Case-controlled Study
Brief Title: Cardiometabolic Care-team Integration Improves Outcomes in Diabetes
Status: Completed | Type: Observational
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Other Study IDs: CEDAR
Record Dates: First submitted 2018-06-02; First posted 2018-06-19 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Cardio-metabolic Care-Team Intervention (CMC-TI)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMC-TI: Cardiometabolic Care Team Intervention
  Interventions: Behavioral: Cardometabolic Team Intervention
- Non-Intervention Comparator site: Non intervention comparator site with usual care

INTERVENTIONS:
Behavioral: Cardometabolic Team Intervention — The CMC-TI team included a registered nurse/certified diabetes educator (RN/CDE) Care Manager, medical assistant (MA) Health Coach, and RN Depression Care Manager. Decision support tools guided therapy for glucose, BP, low-density lipoprotein cholesterol (LDL-c), and depression. At the intervention clinic, the 12-month CMC-TI was delivered to all qualifying patients; surveys were administered to evaluate relevant patient-reported outcomes over 12 months.
  Groups: CMC-TI

SUMMARY:
A pragmatic, quasi-experimental (non-randomized) design was used to evaluate clinical and cost outcomes among patients with type 1 or 2 diabetes (T1D or T2D) at two primary care clinics (n=1 intervention, n=1 usual care) between March 2012 and September 2014. At the intervention clinic, the 12-month Cardio-metabolic Care-Team Intervention (CMC-TI) was delivered to all qualifying patients; surveys were administered to evaluate relevant patient-reported outcomes over 12 months, and a process evaluation gauged CMC-TI feasibility and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 1 and type 2 diabetes

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - All patients with type 1 and type 2 diabetes within two primary care clinics at Scripps Coastal Medical Group.
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 months
  Change in HbA1c between Intervention and Comparator sites

SECONDARY OUTCOMES:
Hospital/ER costs | 12 months
LDL | 12 months
  Change in LDL between Intervention and Comparator sites
Blood pressure | 12 months
  Change in blood pressure between Intervention and Comparator sites

IPD SHARING:
Plan to Share IPD: No